CLINICAL TRIAL: NCT06976164
Title: The Effects of Reflexo Therapy of Sole on Gestational Diabetes Mellitus
Brief Title: Reflexo Therapy for Gestational Diabetes Mellitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Yomna Ghanem, Demonstrator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T. 2024-2025
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Physical Therapy
Keywords: Gestational diabetes mellitus; Foot reflexology; Fasting plasma glucose; 2-h post-prandial glucose; HbA1c
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group A (Experimental)
  Interventions: Procedure: The standard antenatal care.; Procedure: Foot reflexology.
- Experimental Group B (Experimental)
  Interventions: Procedure: The standard antenatal care.

INTERVENTIONS:
Procedure: The standard antenatal care. — Antenatal Protocol.
Procedure: Foot reflexology. — A manual therapy technique.
  Arms: Experimental Group A

SUMMARY:
The purpose of this study will be to detect the effects of Reflexo therapy of sole on GDM.

DETAILED DESCRIPTION:
Gestational diabetes mellitus is considered a hazard factor for antenatal complications for both mother and fetus. It is characterized by glucose intolerance of variable degrees with the beginning or first recognition of pregnancy. It affects 14% of pregnancies worldwide, and it undergoes continuous changes in the diagnostic criteria, ethnicity and the population studied.

There is an increasing prevalence of diabetes mellitus, and its major metabolic disorder caused by the insulin secretion defect or insulin action defect resulting from a defect in insulin secretion, insulin action, or both. As a result, it will lead to chronic hyperglycemia associated with carbohydrates, protein, and fat disturbance.

In spite of the fact that the reason for gestational diabetes mellitus is still not fully understood, it is proposed that human placental lactogen has growth hormone-like actions, and that it causes lipolysis and thus increases the levels of circulating fatty acids that repress the action of insulin and cause insulin resistance in pregnant females which appear to play a crucial role in the pathogenesis of gestational diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. They were maternally aged between 20 and 35 years.
2. The gestational age ranged from between 24 and 36 weeks.
3. Their BMI didn't exceed 30 kg/m2.
4. A singleton live fetus and not under stressful event.

Exclusion Criteria

1. They had high-risk pregnancies.
2. Bad obstetric situations.
3. Diseases that could interfere with participation.
4. Smoking.
5. Oral sedative administration.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 36 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in The Oral Glucose Tolerance Test. | Change from Baseline Oral Glucose Tolerance Test at one month
Change in The Hemoglobin A1C Test. | Change from Baseline Hemoglobin A1C Test at one month

CONTACTS AND LOCATIONS:
Locations (1):
- The Outpatient Clinics, Faculty of Physical Therapy Kafrelsheikh University., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No